CLINICAL TRIAL: NCT04681885
Title: Evaluation of Toothbrush Bristles in Plaque Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CLP-2020-06-01-1
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Plaque, Dental; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Tapered bristles A (Experimental): Test toothbrush with tapered bristle
  Interventions: Device: Tapered bristles A; Device: Tapered bristles B; Device: End rounded bristles
- Tapered bristles B (Active Comparator): Test toothbrush with tapered bristle
  Interventions: Device: Tapered bristles A; Device: Tapered bristles B; Device: End rounded bristles
- End rounded bristles (Active Comparator): Conventionla toothbrush with end rounded bristle
  Interventions: Device: Tapered bristles A; Device: Tapered bristles B; Device: End rounded bristles

INTERVENTIONS:
Device: Tapered bristles A — Subjects use the toothbrush two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week .
Device: Tapered bristles B — Subjects use the toothbrush two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week.
Device: End rounded bristles — Subjects use the toothbrush two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week.

SUMMARY:
The purpose of this cross-over clinical research is to evaluate the cleaning efficacy of toothbrushes tufted with two types of tapered bristles and end rounded bristles in removal of interdental plaque with clinical measurement (Plaque Index) and objective measurement (digitally measured plaque area). This study will demonstrate the influence by a type of processing bristles on removal of interdental plaque and determine an agreement between the different evaluation methods.

This is a randomized evaluator-masked crossover study with 10 subjects. Subjects will be randomly allocated to three test groups. Subjects will use the assigned toothbrush at baseline appointment and two times a day for a week. Plaque Index and plaque area will be assessed before/after one time use at baseline and Day 7. Subjects will be assigned to another toothbrush after one week wash-out period.

ELIGIBILITY:
Inclusion Criteria: Individuals may be included in the study if they meet all of the following inclusion criteria:

* Must have read, understood and signed an informed consent prior to being entered into the study
* Must be 18 to 70 years of age, male or female
* Have at least 20 natural or restored teeth
* Must have average Plaque Index of Ramfjord teeth at baseline greater than 2(Quigley and Hein) at screening
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures (other than those provided during the study) any time during the study
* Agree to refrain from regular oral hygiene regimen for 24 hours and eating for 4 hours before the appointment in the study
* Agree to abstain from the use of any dental products other than those provided in the study
* Agree to comply with the conditions and schedule of the study

Exclusion Criteria: Individuals are not eligible for participation in this study if any of the following are noted:

* Physical limitations or restrictions that might preclude normal tooth brushing
* Evidence of gross oral pathology
* Presence of severe gingivitis with 30 or more sites showing bleeding on probing
* Evidence of major soft tissue lesions or trauma at the baseline visit as determined by the Investigator/Examiner
* Chronic disease with concomitant oral manifestations
* Subjects who are currently undergoing, or require, extensive dental work, orthodontic treatment or periodontal surgery or orthodontic treatment in the preceding 3 months
* Currently using bleaching trays
* Eating disorders
* Recent history of substance abuse
* Smoking >10 cigarettes/day
* Participation in other clinical studies within 14 days of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Garcia-Godoy, DDS, PhD, Principal Investigator — The University of Tennessee Health Science Center
Locations (1):
- The University of Tennessee Health Science Center, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles: Participants were instructed to brush their teeth with test toothbrushes made with following bristles daily for two minutes, using only the provided toothpaste for one-week study period. One-week washout period separates each different intervention of one week.
  First intervention: Tapered bristles A Second intervention: Tapered bristles B Third inetervention: End rounded bristles
- Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A: Participants were instructed to brush their teeth with test toothbrushes made with following bristles daily for two minutes, using only the provided toothpaste for one-week study period. One-week washout period separates each different intervention of one week.
  First intervention: Tapered bristles B Second intervention: End rounded bristles Third inetervention: Tapered bristles A
- End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B: Participants were instructed to brush their teeth with test toothbrushes made with following bristles daily for two minutes, using only the provided toothpaste for one-week study period. One-week washout period separates each different intervention of one week.
  First intervention: End rounded bristles Second intervention: Tapered bristles A Third inetervention: Tapered bristles B
Period: First Intervention (1 Week)
Arm/Group | Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles | Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A | End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles | Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A | End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles | Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A | End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles | Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A | End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Third Intervention (1 Week)
Arm/Group | Tapered Bristles A First, Tapered Bristle B Second, Then End Rounded Bristles | Tapered Bristles B First, End Rounded Bristles Second, Then Tapered Bristles A | End Rounded Bristles First, Tapered Bristles A Second, Then Tapered Bristles B
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Subject disposition for all arms
Arm/Group | Overall Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Navy Plaque Index (Navy Pl) After One-time Brushing
Description: Change of Navy Plaque Index (Navy Pl) after one-time brushing in a whole mouth. The Navy Plaque Index (PI) can be either 0 (plaque is not present) or 1 (plaque is present). Each tooth is partitioned into 9 areas, and the PI is evaluated for teeth numbered 2-15 and 18-31, totaling 28 teeth. Both buccal (B) and lingual (L) sides of each tooth are assessed. The PI value of each person ranges from 0 to 504 (28 teeth × 9 areas × 2 sides). Baseline value is calculated by averaging PI values of 10 subjects before brushing. Post-brushing value is calculated by averaging PI values of 10 subjects after a one-time brushing for 2 minutes
Time Frame: Pre-intervention at baseline and after one-time brushing for 2 minutes at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tapered Bristles A: Subjects use the toothbrush with Tapered bristles A two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method
- Tapered Bristles B: Subjects use the toothbrush with Tapered bristles B two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week.
- End Rounded Bristles: Subjects use the toothbrush with End rounded bristles two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week.
Arm/Group | Tapered Bristles A | Tapered Bristles B | End Rounded Bristles
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Baseline | 367.5 (67.4) | 346.5 (70.4) | 355 (50.9)
  After one-time brushing for 2 minutes | 145.4 (61.8) | 123.8 (59.6) | 130.1 (59.0)

2. Primary Outcome: Change of Digitally Measured Interdental Plaque Area After One-time Brushing
Description: Change of digitally measured interdental plaque area on non-molar teeth, facial/buccal aspect after one-time brushing by image analysis.
Time Frame: Pre-intervention at baseline and after one-time brushing for 2 minutes at baseline
Population: No assessment was done due to: 1. The plaque area is so small as area % in a total region of interest. 2. Regardless of products, most of plaque on teeth surface of buccal side was removed after 2-minute brushing in most of subjects, so it is difficult to detect their difference. 3. Quality of accumulated plaque, e.g. thick but shallow area vs. thin but broad area, is hard to do the assessment. 4. Some photos were not appropriate for image analysis due to being a little out of focus.
Arm/Group | Tapered Bristles A | Tapered Bristles B | End Rounded Bristles
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change of Navy Plaque Index (Navy PI) After 7-day Brushing
Description: Change of Navy Plaque Index (Navy Pl) after 7-day brushing in a whole mouth. The Navy Plaque Index (PI) can be either 0 (plaque is not present) or 1 (plaque is present). Each tooth is partitioned into 9 areas, and the PI is evaluated for teeth numbered 2-15 and 18-31, totaling 28 teeth. Both buccal (B) and lingual (L) sides of each tooth are assessed. The PI value of each person ranges from 0 to 504 (28 teeth × 9 areas × 2 sides). Baseline value is calculated by averaging PI values of 10 subjects before brushing. 7-day value is calculated by averaging PI values of 10 subjects after 7-day brushing.
Time Frame: Pre-intervention at baseline and after 7- day brushing at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tapered Bristles A: Subjects use the toothbrush with two times daily with a fluoride toothpaste for 2 minutes with instructed brushing method for one week .
Arm/Group | Tapered Bristles A | Tapered Bristles B | End Rounded Bristles
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Baseline | 366.3 (67.6) | 346.9 (70.4) | 354.9 (51.2)
  7 days | 372.3 (42.1) | 373.8 (49.8) | 380.1 (44.1)

4. Secondary Outcome: Change of Digitally Measured Interdental Plaque Area After 7-day Brushing
Description: Change of digitally measured interdental plaque area on non-molar teeth, facial/buccal aspect after 7- day brushing by image analysis.
Time Frame: Pre-intervention at baseline and after 7-day brushing at baseline
Population: as for outcome 2
Arm/Group | Tapered Bristles A | Tapered Bristles B | End Rounded Bristles
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 week
Arm/Group | Tapered Bristles A | Tapered Bristles B | End Rounded Bristles
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapered Bristles A (N=10) | Tapered Bristles B (N=10) | End Rounded Bristles (N=10)
Mouth ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Plaque area is not measured by image analysis due to: 1. The plaque area is so small as area% in a total region of interest. 2. Most of plaque on teeth surface of buccal side was removed after 2-minute brushing in most of subjects, so it is difficult to detect their difference. 3. Quality of accumulated plaque, e.g. thick but shallow area vs. thin but broad area, is hard to do the assessment. 4. Some photos were not appropriate for image analysis due to being a little out of focus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04681885/Prot_SAP_000.pdf